CLINICAL TRIAL: NCT03507660
Title: What is the Best Verbal Instruction for Contraction the Pelvic Floor Muscles Among Males
Brief Title: Verbal Instruction for Contraction Pelvic Floor Muscles Among Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Collaborators: Ariel University (Other)
Responsible Party: Principal Investigator, Gali Dar, senior lecturer, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AU-NBA-20180315
Record Dates: First submitted 2018-04-15; First posted 2018-04-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Pelvic Floor Muscle Weakness
Keywords: verbal instruction, pelvic diaphragm, muscle contraction

STUDY DESIGN:
Intervention Model Description: all participants will receive the same six verbal instruction given in a random order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- verbal instruction (Experimental): The participants will be verbal instructed to contract the pelvic floor muscle with the following sentences:
  1. "squeeze the pelvic floor muscles".
  2. "squeeze and lift the pelvic floor muscles as if stopping the flow of urine"
  3. "Take a moderate breath in, let the breath out, draw in and lift your pelvic floor."
  4. ""squeeze the anus"
  5. "shorten the penis"
  6. "elevate the scrotum"
  Interventions: Other: verbal instruction

INTERVENTIONS:
Other: verbal instruction — Verbal instruction for pelvic floor contraction will be given to participants. Ultrasound examination will be conducted to asses urinary bladder displacement being a marker for pelvic floor muscle function.
  Other Names: diagnostic ultrasound assesment

SUMMARY:
The aim of this study is to compare the effectiveness of different verbal instruction on pelvic floor muscle contraction among males. Pelvic floor contraction will be measured via ultrasound.

DETAILED DESCRIPTION:
This study will examine pelvic floor muscle contraction following six different verbal instructions among males. Physical-therapy students will be recruited to complete a survey and non-invasive transabdominal ultrasound assessment.

A bladder filling protocol will be implemented to ensure subjects will have sufficient fluid in their bladders to allow clear ultrasound imaging. This protocol involved subjects consuming 600-750 ml of water in a 1 hr. period. The participants will be tested in a crook-lying supine position with a pillow under their heads for comfort.

All participants will be given six different verbal instructions to contract pelvic floor muscles. Each contraction will be performed 3 time with rests of 10 sec between contractions. While the first 2 contractions for each verbal instruction will be held for 3 sec. the last contraction will be held as long as the participant can conduct and the time of contraction will be measured as well. The pelvic floor contraction will be measured by assessing bladder displacement via diagnostic ultrasound.

To image the pelvic floor a 5 MHz curved linear array transducer (Mindray M5) will be placed in the transverse plane immediately suprapubically over the lower abdomen angled at 15-30 degrees from the vertical. An on screen caliper and measurement tool will be used to measure bladder displacement.

ELIGIBILITY:
Inclusion Criteria:

* willing to participate in the study

Exclusion Criteria:

* none

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — this research will include male population only
Enrollment: 35 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
urinary bladder displacement in millimeters during verbal instructions | up to 6 months
  bladder displacement will be measured via diagnostic ultrasound using the on screen caliper tool

SECONDARY OUTCOMES:
demographic self reported questionnaire regarding height | baseline
  height in meters
demographic self reported questionnaire regarding weight | baseline
  weight in kilograms
self reported questionnaire regarding physical activity | baseline
  number of practice per week
BMI | baseline
  measured in kg/m^2 and calculated from the reported values of weight and height
pelvic floor muscles endurance of contraction in seconds | up to 6 months
  time of muscle contraction will be measured during the last contraction in each instruction
questionnaire regarding symptoms of urinary incontinence = International Consultation on Incontinence Questionnaire - Short Form | baseline
  scale range 0-21 points. higher values represent worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, PHd, Study Director — University of Haifa
Locations (1):
- Ariel University, Department of Physical Therapy, Ariel, Israel

IPD SHARING:
Plan to Share IPD: Yes
The result of the study will be analysed. a paper will be submitted to international journal with study description including methods, examination protocol results.
Supporting Information: Study Protocol, CSR
Time Frame: The result of the study will be analysed. a paper will be submitted to international journal with study description including methods, examination protocol results.
Access Criteria: according to journal policy

REFERENCES:
- [Result] Stafford RE, Coughlin G, Lutton NJ, Hodges PW. Validity of Estimation of Pelvic Floor Muscle Activity from Transperineal Ultrasound Imaging in Men. PLoS One. 2015 Dec 7;10(12):e0144342. doi: 10.1371/journal.pone.0144342. eCollection 2015. PMID 26642347